CLINICAL TRIAL: NCT02587468
Title: Bioavailability and Absorption Kinetics of Phenolic Compounds and Specific Vitamins of a Commercially Available, Encapsulated Nutraceutical (Juice Plus+®)
Brief Title: Bioavailability and Absorption Kinetics of Phenolic Compounds and Specific Vitamins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Beat (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Principal Investigator, Green Beat
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 27-507 ex 14/15
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: phenolics; absorption; fruit & vegetable concentrate; Bioavailability of phenolic compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Juice Plus+(R) (Experimental): Check of phenolic absorption between baseline and after 8wks of intake before-after comparison
  Interventions: Dietary Supplement: Juice Plus+(R)

INTERVENTIONS:
Dietary Supplement: Juice Plus+(R) — before-after comparison of plasma phenolics

SUMMARY:
GOAL To identify absorption kinetics and bioavailability of phenolic compounds and specific vitamins from encapsulated Juice Plus+® powder

ENDPOINTS

* Absorption kinetics of phenolic compounds in plasma
* Bioavailability of vitamins C, E, and carotenoids into plasma

Subjects: 20 healthy subjects from Graz region, meeting all inclusion criterions (see underneath).

DETAILED DESCRIPTION:
Phytonutrients are regarded to play an important role in many health-related issues like:

* Improvement of redox balance
* Anti-inflammatory effects
* Prevention of chronic diseases like CVD, stroke, diabetes II, Alzheimer´s, AMD, and certain forms of cancer
* Beneficial effects on human´s microbiome Therefore it is of scientific interest whether this product provides absorbable phytonutrients/phenolics and vitamins to support mechanistic explanations for the beneficial outcomes observed in the past after intake of Juice Plus+®.

GOAL To identify absorption kinetics and bioavailability of phenolic compounds and specific vitamins from encapsulated Juice Plus+® powder

MERITS

* This study would reveal knowledge whether and to which extent specific vitamins and phenolic compounds are absorbed, including absorption kinetics/metabolism.
* Data of this study may provide support for mechanistic arguments on the beneficial clinical outcomes observed and published in the past.

ENDPOINTS

* Absorption kinetics of phenolic compounds in plasma
* Bioavailability of vitamins C, E, and carotenoids into plasma

Absorption kinetics of phytonutrients:

* Open-, one-arm study, absorption kinetics over 10 hours
* 5 blood sample collections: baseline (= 0); 1hr, 2hrs, 5hrs and 10 hours after intake of 3 capsules
* Wash-out of all food supplements and dietetic foodstuff: 2 weeks
* Wash-out of phytonutrients: 48 hours before baseline sampling, accomplished via a phytonutrient-poor diet.

Bioavailability of vitamins C, E, A and carotenoids:

* Open-, one-arm study over 8 weeks
* 2 blood sample collections: at baseline (2 weeks after the phenolics experiment) and after 8-weeks
* Wash-out of all food supplements and dietetic foodstuff: 4 weeks, 2 weeks before the phenolics experiment + another 2 weeks Subjects: 20 healthy subjects from Graz region, meeting all inclusion criterions (see underneath).

ELIGIBILITY:
Inclusion Criteria:

* 20 healthy men and women, 20-50 years old;
* non-smokers;
* BMI >20 und <30 kg/m2;
* no medication;
* premenopausal;
* normal dietary habits (no specific diets, meals, food components etc.);
* adherence to wash-out period.

Exclusion Criteria:

* all people not meeting the inclusion criterions;
* diet: subjects consuming >4 servings of fruits and vegetables per day;
* subjects with any kind of food allergy or histamine intolerance;
* highly trained subjects (> 5 training units/week);
* women with menstrual dysfunctions;
* pregnancy
* alcoholics.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Absorption kinetics of phenolic acids after 1, 2, 5 and 10 hours, measured via HPLC, evaluated by repeated measures ANOVA, and assessed via SPSS 19.0. | 1 year
  For the phenolics analyses subjects come to the lab after an overnight fast, and after 2 weeks wash-out of all food supplements and 48 hours wash-out of phytonutrients (phytonutrient-poor diet). To adhere to the phytonutrient-poor diet they receive an exact diet plan in the forefront. This plan will be perused with the research associate. After the baseline blood drawing, they receive 3 capsules of Juice Plus+® consumed with 250ml plain water from the pipe. They will be instructed to swallow one capsule of each blend (fruit, berry, vegetable). During this day 4 additional blood samples will be drawn: 1hr, 2hrs, 5hrs, 10hrs after capsule intake in the morning.
  After the 2hrs blood sampling the subjects get a standardized, phytonutrient-poor snack: white bread, cheese, ham, milk and water ad libitum. Subjects will receive a list with suggestions of allowed food they could consume on this day.

SECONDARY OUTCOMES:
Absorption of ß-carotene after 8 weeks of supplementation, measured via HPLC, evaluated by paired t-test, and assessed via SPSS 19.0 | 1 year
  Two weeks after the first blood drawings, for the phytonutrient absorption and absorption kinetics, subjects will be invited to another visit to the laboratory. During these two weeks the volunteers adhere to the wash-out from all food supplements. After an overnight fast they come to the lab for the baseline blood drawings to evaluate vitamins and carotenoids absorption. This procedure will be repeated after 8 weeks of supplementation with 6 capsules of Juice Plus+® per day (~2.2g juice powder per day). During this time subjects will be instructed to maintain their habitual diet.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, PhD, Principal Investigator — Green Beat + Medical University of Graz
Locations (2):
- Austria (2):
  - Institute of Pathophysiology and Immunology, Graz, Styria
  - Green Beat, Graz